CLINICAL TRIAL: NCT03702530
Title: Immunisation, Treatment and Controlled Human Hookworm Infection
Acronym: ITCHHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ITCHHI
Record Dates: First submitted 2018-08-10; First posted 2018-10-11 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Necator Americanus Infection

STUDY DESIGN:
Intervention Model Description: Volunteers are randomized into either the intervention or the placebo group (2:1 allocation). The two groups run parallel in the trial. At the moments of immunization in the intervention group volunteers in the placebo group receive a mock infection with water to maintain blinding.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, clinical trial physicians and laboratory personnel are blinded for treatment allocation. Blinding is maintained by exposing the volunteers in the placebo group to a mock infection with water. During the trial clinical trial physicians are blinded to the outcome measures (i.e. Kato-Katz outcomes), laboratory staff are blinded for the study code of samples delivered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 3x 50 L3 larvae immunisation with albendazole treatment and 2x 50 L3 larvae infection
  Interventions: Biological: 3x 50 L3 larvae immunisation with albendazole treatment; Biological: 2x 50 L3 larvae infection
- Placebo (Placebo Comparator): 3x placebo immunisation with albendazole treatment and 2x 50 L3 larvae infection
  Interventions: Other: 3x placebo immunisation with albendazole treatment; Biological: 2x 50 L3 larvae infection

INTERVENTIONS:
Biological: 3x 50 L3 larvae immunisation with albendazole treatment — Immunisation with 50 Necator americanus L3 larvae at week 0, 3 and 6 with albendazole treatment at week 2, 5 and 8
  Arms: Intervention
Other: 3x placebo immunisation with albendazole treatment — Mock immunisation with water at week 0, 3 and 6 with albendazole treatment at week 2, 5 and 8
  Arms: Placebo
Biological: 2x 50 L3 larvae infection — After (mock) immunisation, infection with 50 Necator americanus larvae at week 13 and 15

SUMMARY:
24 healthy volunteers will be immunized with three times 50 L3 larvae or placebo followed by treatment with albendazol and subsequently challenged with twice 50 L3 larvae.

DETAILED DESCRIPTION:
24 healthy hookworm-naive volunteers will be randomized in a 2:1 allocation to either the intervention group or placebo. Volunteers in the intervention group will be immunized three times with 50 L3 larvae of Necator americanus with three-week intervals. Two weeks after each immunization, volunteers will be treated with albendazole. Four weeks after the last treatment all volunteers are challenged with controlled human hookworm infection consisting of two doses of 50 L3 larvae with a two week interval. 16 weeks after the first challenge all volunteers will be treated with albendazole, except up to four volunteers who will be asked to remain as chronic donors for future hookworm studies.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Subject is aged ≥ 18 and ≤ 45 years and in good health.
2. Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
3. Subject is able to communicate well with the investigator and is available to attend all study visits.
4. Subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period.
5. For female subjects: subject agrees to use adequate contraception and not to breastfeed for the duration of study.
6. Subject agrees to refrain from travel to a hookworm endemic area during the course of the trial.
7. Subject has signed informed consent.

Exclusion Criteria:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immune-deficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following:

   * positive HIV, HBV or HCV screening tests;
   * the use of immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period;
   * having one of the following laboratory abnormalities: ferritine <10 ug/L, transferrine <2.04 g/L or Hb <6.5 mmol/L for females or <7.5 mmol/L for males.
   * history of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years;
   * any history of treatment for severe psychiatric disease by a psychiatrist in the past year;
   * history of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset;
   * inflammmatory bowel syndrome;
   * regular constipation, resulting in bowel movements less than three times per week.
2. Known hypersensitivity to or contra-indications for use of albendazole, including co-medication known to interact with albendazole metabolism (e.g. carbamazepine, phenobarbital, phenytoin, cimetidine, theophylline, dexamethasone).
3. Known allergy to amphotericin B or gentamicin.
4. For female subjects: positive urine pregnancy test at screening.
5. Positive faecal qPCR for hookworm at screening, any known history of hookworm infection or treatment for hookworm infection.
6. Being an employee or student of the department of Parasitology of the LUMC.
7. Current or past scars, tattoos, or other disruptions of skin integrity at the intended site of larval application.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Difference between egg counts between intervention and placebo group | week 25-29
  Comparison of average egg counts from week 25-29 of the trial (which is week 12 to 16 after controlled human hookworm infection) by Kato-Katz between intervention group and placebo group

SECONDARY OUTCOMES:
Frequency of adverse events | week 0-29
  Comparison of frequency of adverse events collected during immunisation phase and after controlled human hookworm infection between intervention and placebo group
Severity of adverse events | week 0-29
  Comparison of severity of adverse events collected during immunisation phase and after controlled human hookworm infection between intervention and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: M. Roestenberg, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoogerwerf MA, Janse JJ, Kuiper VP, van Schuijlenburg R, Kruize YC, Sijtsma JC, Nosoh BA, Koopman JR, Verbeek-Menken PH, Westra IM, Meij P, Brienen EA, Visser LG, van Lieshout L, Jochems SP, Yazdanbakhsh M, Roestenberg M. Protective efficacy of short-term infection with Necator americanus hookworm larvae in healthy volunteers in the Netherlands: a single-centre, placebo-controlled, randomised, controlled, phase 1 trial. Lancet Microbe. 2023 Dec;4(12):e1024-e1034. doi: 10.1016/S2666-5247(23)00218-5. PMID 38042152